CLINICAL TRIAL: NCT03358576
Title: Prospective, Phase 3, Randomized, Multi-center, Double-blind Study of Efiicacy, Tolerability & Safety of Sulopenem & Sulopenem-etzadroxil/Probenecid vs Ertapenem Followed by Cipro-metronidazole for Treatment of cIAI in Adults
Brief Title: Sulopenem Versus Ertapenem for Complicated Intra-abdominal Infection (cIAI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT001-303
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2019-11

CONDITIONS: Intra Abdominal Infections
MeSH Terms: conditions — Intraabdominal Infections | interventions — Ertapenem; Probenecid; Ciprofloxacin; Metronidazole; Amoxicillin-Potassium Clavulanate Combination; sulopenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulopenem (Experimental): Sulopenem 1000 mg IV once daily for at least 5 days, followed by Sulopenem-Etzadroxil/Probenecid 500 mg PO twice daily to complete 7-10 days of treatment
  Interventions: Drug: Sulopenem-Etzadroxil/Probenecid; Drug: Sulopenem
- Ertapenem (Active Comparator): Ertapenem 1000 mg IV once daily for at least 5 days, followed by ciprofloxacin 500 mg PO twice daily along with metronidazole 500 mg PO four times daily. If patient is found to have causative pathogens that are resistant to ciprofloxacin they will receive amoxicillin-clavulanate 875 mg PO twice daily instead
  Interventions: Drug: Ertapenem; Drug: Ciprofloxacin; Drug: Metronidazole; Drug: Amoxicillin-Clavulanate

INTERVENTIONS:
Drug: Ertapenem — Antibiotic for complicated intra-abdominal infection
  Other Names: Invanz
  Arms: Ertapenem
Drug: Sulopenem-Etzadroxil/Probenecid — Antibiotic for complicated intra-abdominal infection
  Arms: Sulopenem
Drug: Ciprofloxacin — Antibiotic for complicated intra-abdominal infection
  Other Names: Cipro
  Arms: Ertapenem
Drug: Metronidazole — Antibiotic for complicated intra-abdominal infection
  Other Names: Flagyl
  Arms: Ertapenem
Drug: Amoxicillin-Clavulanate — Antibiotic for complicated intra-abdominal infection
  Other Names: Augmentin
  Arms: Ertapenem
Drug: Sulopenem — Antibiotic for complicated intra-abdominal infection
  Arms: Sulopenem

SUMMARY:
This is a prospective, Phase 3, randomized, multi-center, double-blind study of the efficacy, tolerability and safety of sulopenem followed by sulopenem-etzadroxil/probenecid versus ertapenem followed by ciprofloxacin-metronidazole for treatment of complicated intra-abdominal infections in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or the patient's legally acceptable representative able to provide a signed written informed consent prior to any study-specific procedures.
2. Adult patients ≥18 years of age
3. EITHER:

   a. Intra-operative/post-operative enrollment with visual confirmation (presence of pus within the abdominal cavity) of an intra-abdominal infection associated with peritonitis including at least 1 of the following diagnosed during the surgical intervention: i. Cholecystitis with gangrenous rupture or perforation or progression of the infection beyond the gallbladder wall ii. Diverticular disease with perforation or abscess iii. Appendiceal perforation or peri-appendiceal abscess iv. Traumatic perforation of the intestines, only if operated on >12 hours after perforation occurs v. Secondary peritonitis (but not spontaneous bacterial peritonitis associated with cirrhosis and chronic ascites) vi. Intra-abdominal abscess (including of liver or spleen provided that there was extension beyond the organ with evidence of intraperitoneal involvement).

   OR:

   b. Pre-operative enrollment where one of the following surgical procedures are planned within 24 hours prior to the first dose of study drug: i. Open laparotomy, percutaneous drainage of an intra-abdominal abscess, or laparoscopic surgery.
4. Evidence of systemic inflammatory indicators, with at least one of the following:

   i. Fever (defined as body temperature >38°C) or hypothermia with a core body temperature <35°C ii. Elevated white blood cell count (>12,000 cells/mm3) iii. Drop in blood pressure (systolic BP must be <90 mmHg without pressor support) iv. Increased heart rate (>90 bpm) and respiratory rate (>20 breaths/min) v. Hypoxia (oxygen saturation ≤90 percent on room air)
5. Physical findings or symptoms consistent with intra-abdominal infection, with at least one of the following:

   i. Abdominal pain and/or tenderness, with or without rebound ii. Localized or diffuse abdominal wall rigidity iii. Abdominal mass iv. Nausea/vomiting v. Altered Mental Status
6. Specimen/s from the surgical intervention were sent for culture.

Exclusion Criteria:

1. Patient diagnosed with traumatic bowel perforation undergoing surgery within 12 hours; perforation of gastroduodenal ulcers undergoing surgery within 24 hours. Other intra-abdominal processes in which the primary etiology was not likely to be infectious.
2. Patient has abdominal wall abscess or bowel obstruction without perforation or ischemic bowel without perforation.
3. Patient has simple cholecystitis or gangrenous cholecystitis without rupture, or simple appendicitis, or acute suppurative cholangitis; or infected necrotizing pancreatitis or pancreatic abscess.
4. Patient whose surgery included staged abdominal repair, or "open abdomen" technique, or marsupialization.
5. Patient known at study entry to have a complicated intra-abdominal infection caused by pathogens resistant to the study antimicrobial agents.
6. Patient needed effective concomitant systemic antibacterials (oral, IV, or intramuscular) or antifungals in addition to those designated in the 2 study groups, except vancomycin, linezolid, or daptomycin if started for known or suspected methicillin-resistant Staphylococcus aureus (MRSA) or Enterococcus spp. as per clinical study protocol (CSP).
7. Patient has perinephric infections or an indwelling peritoneal dialysis catheter.
8. Patient has suspected intra-abdominal infections due to fungus, parasites (e.g., amoebic liver abscess), virus, or tuberculosis.
9. Patient has a known history of serious allergy, hypersensitivity or any serious reaction to carbapenem antibiotics, or to other β-lactam antibiotics
10. Patient known to have any of the following laboratory values as defined below:

    1. Hematocrit <25% or hemoglobin <8 g/dL
    2. Absolute neutrophil count <1000/mm3
    3. Platelet count <75,000/mm3
    4. Bilirubin >3 x the upper limit of normal (ULN), unless isolated hyperbilirubinemia was directly related to the acute infection or known Gilbert's disease
    5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 x ULN values at Screening. Patients with elevations of AST and/or ALT up to 5 x ULN will be eligible if these elevations are acute and directly related to the infectious process being treated. This must be documented
    6. Alkaline phosphatase (ALP) >3 x ULN. Patients with values >3.0 x ULN and <5.0 x ULN are eligible if this value is acute and directly related to the infectious process being treated. This must be documented.
    7. Estimated creeatinine clearance <50 mL/min
11. Patient has a body mass index >45 kg/m2.
12. Patient has APACHE II score >30.
13. Patient considered unlikely to survive the 4-week study period or has a rapidly progressive or terminal illness, including septic shock that was associated with a high risk of mortality.
14. Patient unlikely to respond to 10-14 days of treatment with antibiotics.
15. Patient received systemic antibacterial agents within the 72-hour period prior to study entry, unless either of the following pertained:

    a. Patient has a new infection (not considered a treatment failure) and both of the following were met: i. Patient received no more than 24 hours of total prior antibiotic therapy ii. Patient received ≤1 dose of a treatment regimen post-operatively and antibiotics were not received more than 6 hours post-procedure.

    b. Patient considered to have failed the previous treatment regimen i.e., pre-operative treatment of any duration with non-study systemic antimicrobial therapy for peritonitis or abscess permitted provided that all of the following are met: i. The treatment regimen had been administered for at least 72 hours and was judged to have been inadequate ii. The patient had an operative intervention that was just completed or was intended no more than 24 hours after study entry iii. Findings of infection were documented at surgery iv. Specimens for bacterial cultures and susceptibility testing were taken at operative intervention v. No further non-study antibacterials were administered after randomization.
16. Patient has a concurrent infection that may interfere with the evaluation of response to the study antibiotic.
17. Patient receiving hemodialysis or peritoneal dialysis.
18. Patient has a history of acute hepatitis in the recent past (3 months prior to study entry), chronic hepatitis, cirrhosis, acute hepatic failure, or acute decompensation of chronic hepatic failure.
19. Patient has past or current history of epilepsy or seizure disorders excluding febrile seizures of childhood.
20. Patient immunocompromised as evidenced by any of the following:

    1. Human immunodeficiency virus infection, with either a recent (in the past 6 months) acquired immune deficiency syndrome-defining condition or a CD4 + T lymphocyte count <200/mm3
    2. Systemic or hematological malignancy requiring chemotherapeutic or radiologic/immunologic interventions within 6 weeks prior to randomization, or anticipated to begin prior to completion of study
    3. Immunosuppressive therapy, including maintenance corticosteroid therapy (>40 mg/day equivalent prednisolone) for 5 days or more.
21. Patient participating in any other clinical study that involved the administration of an investigational medication at the time of presentation, during the course of the study, or who had received treatment with an investigational medication in the 30 days prior to study enrollment, or had previously been enrolled in this study or had been treated with sulopenem.
22. Patient is in a situation or has a condition that, in the investigator's opinion, may interfere with optimal participation in the study.
23. Patient unlikely to comply with protocol e.g., uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.
24. Patient has known inflammatory bowel disease (ulcerative colitis or Crohn's disease) or Clostridium difficile-associated diarrhea.
25. Patients with a history of blood dyscrasias
26. Patients with a history of uric acid kidney stones
27. Patients with acute gouty attack
28. Patients on chronic methotrexate therapy
29. Females of child-bearing potential who are unable to take adequate contraceptive precautions, have a positive pregnancy test result within 24 hours of study entry, are otherwise known to be pregnant, or are currently breastfeeding an infant.
30. Male subjects who do not agree to use an effective barrier method of contraception during the study and for 14 days post treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (11):
  - Medical Facility, Chula Vista, California
  - Medical Facility, Torrance, California
  - Medical Facility, Idaho Falls, Idaho
  - Medical Facility, Boston, Massachusetts
  - Medical Facility, Royal Oak, Michigan
  - Medical Facility, St Louis, Missouri
  - Medical Facility, Butte, Montana
  - Medical Facility, Lincoln, Nebraska
  - Medical Facility, Omaha, Nebraska
  - Medical Facility, Somers Point, New Jersey
  - Medical Facility, Columbus, Ohio
- Bulgaria (7):
  - Medical Facility, Blagoevgrad
  - Medical Facility, Lom
  - Medical Facility, Pleven
  - Medical Facility, Plovdiv
  - Medical Facility, Rousse
  - Medical Facility, Sofia
  - Medical Facility, Varna
- Estonia (5):
  - Medical Facility, Kohtla-Järve
  - Medical Facility, Tallinn
  - Medical Facility, Tartu
  - Medical Facility, Viljandi
  - Medical Facility, Võru
- Georgia (3):
  - Medical Facility, Gori
  - Medical Facility, Kutaisi
  - Medical Facility, Tbilisi
- Hungary (3):
  - Medical Facility, Kaposvár
  - Medical Facility, Pécs
  - Medical Facility, Veszprém
- Latvia (3):
  - Medical Facility, Daugavpils
  - Medical Facility, Rēzekne
  - Medical Facility, Riga
- Medical Facility, Bielsk Podlaski, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulopenem | Ertapenem
Started | 338 | 336
Completed | 312 | 311
Not Completed | 26 | 25

BASELINE CHARACTERISTICS:
Population: complicated intra-abdominal infections
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulopenem | Ertapenem | Total
Number analyzed (Participants) | 338 | 336 | 674
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 226 | 217 | 443
  >=65 years | 112 | 119 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (18.4) | 54.8 (18.0) | 54.3 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 155 | 315
  Male | 178 | 181 | 359
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 329 | 328 | 657
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Latvia | 26 | 30 | 56
  Hungary | 25 | 21 | 46
  United States | 16 | 16 | 32
  Georgia | 38 | 45 | 83
  Estonia | 37 | 40 | 77
  Czechia | 10 | 7 | 17
  Russia | 19 | 21 | 40
  Serbia | 5 | 12 | 17
  Ukraine | 64 | 54 | 118
  Bulgaria | 98 | 90 | 188
creatinine clearance [Mean (Standard Deviation); unit: mL/min] | 92.7 (41.4) | 87.9 (39.1) | 90.3 (87.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Success
Description: Clinical response is defined as resolution in signs and symptoms of the index infection and no new symptoms, without the need for additional antibiotics or interventions
Time Frame: Day 28 +/- 1 day
Population: micro-MITT population
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem | Ertapenem
Number analyzed (Participants) | 249 | 266
percentage of participants | 85.5 | 90.2

2. Secondary Outcome: Percentage of Participants With Clinical Success
Description: as for outcome 1
Time Frame: Day 11-14 +/- 1 day
Population: micro-MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem | Ertapenem
Number analyzed (Participants) | 249 | 266
Participants | 208 | 227

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the test-of-cure visit, an average of 28 days
Arm/Group | Sulopenem | Ertapenem
All-Cause Mortality (participants affected / at risk) | 4/338 | 4/336
Serious Adverse Events (participants affected / at risk) | 25/338 | 12/336
Other Adverse Events (participants affected / at risk) | 0/335 | 0/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulopenem (N=338) | Ertapenem (N=336)
Abdominal abscess (Infections and infestations) | 6 (6) | 0 (0)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
small intestine obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
pyrexia (General disorders) | 1 (1) | 0 (0)
sudden death (General disorders) | 1 (1) | 0 (0)
systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
liver abscess (Infections and infestations) | 2 (2) | 1 (1)
appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
colon gangrene (Infections and infestations) | 1 (1) | 0 (0)
peritonitis (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
internal hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide manuscripts, abstracts, or full text of any other intended disclosure (poster, invited speaker or guest lecturer, etc) to Iterum at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, the PI agrees to delay disclosure for a period not to exceed an additional 60 days. The PI will, on request, remove any previously undisclosed Confidential Information before disclosure.

DOCUMENTS (2):
  • Study Protocol (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03358576/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT03358576/SAP_001.pdf